CLINICAL TRIAL: NCT05152212
Title: An Open Label, Phase I Trial of LVGN7409 as Single Agent in Locally Advanced, Metastatic or Recurrent/Refractory Malignancy
Brief Title: Study of LVGN7409 (CD40 Agonist Antibody) in Locally Advanced, Metastatic or Recurrent/Refractory Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lyvgen Biopharma Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVGN7409-201
Record Dates: First submitted 2021-11-09; First posted 2021-12-09 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LVGN7409 (Experimental): Monotherapy Dose Escalation
  Interventions: Biological: LVGN7409

INTERVENTIONS:
Biological: LVGN7409 — Route of administration is IV infusion, and the frequency of administration is once every 3 weeks(Q3W). One cycle is 3 weeks, and treatment can be up to 35 cycles if patients receive benefits.

SUMMARY:
The study of LVGN7409-201 is designed to use a bridging dose escalation to quickly establish the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE) as well as the recommended Phase 2 dose(s) (RP2D) of LVGN7409 as a single agent (monotherapy) in the treatment of locally advanced, metastatic or recurrent/refractory malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years.
* Ability to understand and willingness to sign a written informed consent document (ICF).
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* Estimated life expectancy, in the judgment of the Investigator, of at least 90 days.
* Adequate bone marrow function, as defined by all of the following:

  1. hemoglobin (Hb) ≥ 9.0 g/dL, and
  2. absolute neutrophil count (ANC) ≥ 1.5x10 9/L, and
  3. platelet count (PLT) ≥ 75x10 9/L.
* Adequate liver function, as defined by all of the following:

  1. Total bilirubin ≤ 1.5 × ULN; or ≤ 2.5 × ULN for patients who have serum bilirubin increases due to underlying Gilbert's Syndrome or familial benign unconjugated hyperbilirubinemia.
  2. Aspartate Aminotransferase (AST) ≤ 1.5 × ULN, and Alanine Transaminase (ALT) ≤ 1.5× ULN.
  3. International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT)- ≤1.5 × ULN unless participant is receiving anticoagulant therapy and levels are within the therapeutic range.
  4. Amylase and lipase ≤1.5 × ULN
* Adequate renal function as defined by an estimated serum creatinine clearance of ≥ 50 mL/min (calculated by Cockcroft-Gault formula) .
* Women of childbearing potential must agree to abstain from heterosexual intercourse or use highly effective contraceptive methods from the time of signing informed consent and through 120 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she (or her partner) is participating in this study, she should inform her treating physician immediately.

  a. A woman of childbearing potential is any woman, regardless of sexual orientation, who meets the following criteria: 1. has not undergone tubal ligation, a hysterectomy, or bilateral oophorectomy; or 2. has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Men enrolled on this study must agree to abstain, be surgically sterilized, or agree to use highly effective methods of contraception, including barrier contraception from the time of signing informed consent and through 120 days after the last dose of study drug.
* Patients should recover from all reversible clinically significant AEs of previous anticancer therapies to baseline or NCI-CTCAE v. 5.0 Grade 0-1, except for alopecia (any Grade), Grade < 2 sensory or motor peripheral neuropathy, lymphopenia, or hypothyroidism on hormone replacement (Grade 2), within 14 days prior to the first dose on study. Inclusion of patients with other toxicities deemed not clinically significant (Grade ≤ 2) should be discussed and approved by the Medical Head of Sponsor.
* Patients infected with the HIV virus will be eligible if their CD4 count is > 350 cells/ μL or if they have no history of AIDS defining infections within the past 12 months. Trial participants should be on anti-retroviral therapy for at least 4 weeks and have an HIV viral load < 400 copies/mL.
* All acute adverse reactions caused by previous anti-tumor treatment or surgery were alleviated to a satisfactory level.

Addtional inclusion criteria of Phase Ia:

* Histologically/cytologically confirmed, locally advanced relapsed, unresectable or metastatic solid tumors and lymphomas that are refractory or intolerant to standard of care therapy, or for which no standard therapy exists.

Addtional inclusion criteria of Phase Ib:

* All patients in Phase 1b must have at least one measurable lesion as defined by RECIST v1.1 for solid tumors.

Note: Tumor lesions that are situated in a previously irradiated area will be considered measurable, provided sufficient time has elapsed to demonstrate a response (if any) followed by clear imaging-based progression of the lesions since the time of radiation.

* All patients in Phase 1b with advanced/metastatic malignancy receiving LVGN7409 as monotherapy must have received one prior line of approved therapy, such as treatment with or without immune checkpoint inhibitor and with documented progression or relapse or intolerable.

Exclusion Criteria:

* Prior therapy with anti-CD40 therapy including Bispecific antibody.
* Receipt of systemic anticancer therapy including investigational agents or devices within 5 half-lives of the first dose of study treatment. For anticancer therapies with half-life greater than 5 days, a washout of 21 days or longer is acceptable
* The subject was experienced radiotherapy within 14 days before the first dose of study treatment. [Previous radiotherapy to the central nervous system (CNS) within 28 days of the first dose of study treatment].
* Prior exposure to immune-therapeutics is allowed, including PD-1 and PD-L1 inhibitors, provided the participant did not experience Grade ≥ 3 drug-related toxicity, or a toxicity requiring discontinuation of the PD-1 or PD-L1 inhibitor.
* Known unstable CNS metastasis and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically and radiographically stable, without evidence of recurrence/progression, have no evidence of new or enlarging brain metastases or encephaledema, and are using no corticosteroids for at least 7 days prior to study medication.
* Received a live-virus vaccine within 30 days of the first dose of study drug.
* Grade ≥ 3 allergic reaction to treatment with a monoclonal antibody or has a known or suspected hypersensitivity to components of the study treatment(s).
* Baseline QT interval corrected by Fridericia's formula (QTcF) > 480 milliseconds or known to have congenital prolonged QT syndrome.
* History of Grade ≥ 3 immune-related AEs (irAEs). Exceptions: hypothyroidism, type 1 diabetes mellitus (Type 1 DM), and dermatologic irAEs (patients with previous Steven Johnson Syndrome, toxic epidermal necrolysis or other severe forms of dermatitis are ineligible) are allowed. Type 1 DM should be controlled with HbA1c <8% as per ADA recommendation.
* Receiving an immunologically based treatment for any reason, including chronic use of systemic steroids equivalent to > 10 mg/day of prednisone within 7 days of the first dose of study drug or at any time during study participation.

Note: Use of inhaled or topical steroids or systemic corticosteroids equivalent to ≤ 10 mg/day prednisone equivalent is permitted as is short-term use of corticosteroids at doses equivalent to > 10 mg/day of prednisone (e.g., pre-medication prior to contrast).

* Treatment with systemic immune-stimulatory agents (e.g., IL-2, IFNγ) within 4 weeks prior to the first dose of study drug.
* History or current active or chronic autoimmune disease including but not limited to inflammatory bowel disease, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease.

(Exception: Patients with vitiligo or resolved childhood asthma/atopy, hypothyroidism on stable hormone replacement, controlled asthma, Type I diabetes, Graves' disease, Hashimoto's disease, or with Medical Monitor approval)

* Clinically significant cardiac condition, including unstable angina, acute myocardial infarction within 6 months of Cycle 1 Day 1, New York Heart Association Class III or IV congestive heart failure, unstable angina pectoris or arrhythmia requiring therapy.

Note: A patient with an arrhythmia may enroll if the patient is on antiarrhythmic medication and is in a rate- controlled rhythm on the screening electrocardiogram (ECG).

* Pleural effusion or pericardial effusion with uncontrolled or requiring repeat drainage (recurrence within two weeks after intervention), or recurrent ascites requiring drainage ≥ once a month.
* Active infection requiring intravenous (IV) anti-infectives within 14 days before the first dose of study treatment, or nonhealing wound or ulcer.
* Current evidence or history of interstitial lung disease or active, noninfectious pneumonitis requiring treatment such as oral or intravenous glucocorticoids.
* Female patients who are pregnant or breastfeeding (confirmation that the patient is not pregnant must be by a negative serum pregnancy test result obtained during screening; pregnancy testing is required of women of childbearing potential but not required for postmenopausal or surgically sterilized women), or expecting to conceive children within the duration of the study, beginning at the screening visit (Initial Visit) through 120 days after the last dose of study treatment.
* Any evidence of severe or uncontrolled systemic disease including, but not limited to, active bleeding diathesis, organ transplantation, or active COVID-19 infection with a detectable viral load.
* Any evidence of severe or uncontrolled systemic disease including, but not limited to, active bleeding diathesis, organ transplantation, or active COVID-19 infection with a detectable viral load.
* Subjects with known positive test results of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illnesses/conditions, which in the judgment of the Investigator might compromise the safety of the patient, integrity of the study, interfere with the patient participation in the study, or compromise the study objectives.
* Previously received an allogeneic tissue/organ transplant, stem cell or bone marrow transplant or solid organ transplant.
* History of Car-T therapy.
* History of hemorrhagic or ischemic stroke within the last 6 months.
* History of malignancy within the previous 2 years except for localized cancers that are not related to the current cancer being treated, are considered to have been cured and in the opinion of the Investigator, present a low risk for recurrence, including basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
MTD and/or RDE and RP2D | up to 24 months
  MTD or RDE or RP2D will be determined according to safety, tolerability, Pharmacokinetic (PK) profile and clinical activity.
Incidence rate of Dose-limiting Toxicity (DLT) within 3 weeks after first dose | up to 24 months
  Incidence rate of dose-limiting toxicities within 3 weeks after first dose
Safety and tolerability (Serious adverse events, adverse events, dose-limiting toxicities, Maximum Tolerated Dose) | up to 24 months
  Adverse events will be assessed, and severity will be assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (ECI CTCAE) v5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  ORR will be documented as the percentage of paritcipants who achived either complete response (CR) or partial response (PR), as assessed based on RECIST v1.1 and iRECIST critieria.
Disease Control Rate (DCR) | up to 24 months
  DCR will be documented as the percentage of participants who achived CR, PR or stable disease (SD), as assessed based on RECIST v1.1 and iRECIST critieria.
Duration of Respons (DOR) | up to 24 months
  DOR will be documented as the time from the date on which objective response (CR or PR).
PK parameter | up to 24 months
  PK parameter：AUC0-∞
PK parameter | up to 24 months
  PK parameter：AUC0-t
PK parameter | up to 24 months
  PK parameter：Cmax
PK parameter | up to 24 months
  PK parameter：Tmax
PK parameter | up to 24 months
  PK parameter：T1/2
PK parameter | up to 24 months
  PK parameter：CL
Anti drug antibody (ADA) to LVGN7409 | up to 24 months
  The presence of ADA directed against LVGN7409 will be determined.

OTHER OUTCOMES:
Biomarkers PD-L1/ MSI/dMMR and/or tumor mutational burden (TMB) | up to 24 months
  Level of PD-L1/ MSI/dMMR and/or TMB will be assessed.
Biomarkers IL-6, IL-12, TNF-α, IFN-γ and soluble CD40 antigen | up to 24 months
  Level of IL-6, IL-12, TNF-α, IFN-γ and soluble CD40 antigen in serum will be assessed.
Immune cell typing in peripheral blood, CD40 receptor occupation in B lymphocyte cell. | up to 24 months
  The change of biomarkers will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Center Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China